CLINICAL TRIAL: NCT06978751
Title: Development of a Risk Assessment Tool for Incontinence-associated Dermatitis (IAD): a Cohort Study on the Predictive Performance of Risk Factors for IAD
Acronym: INCONTECT
Status: Enrolling by invitation | Type: Observational
Sponsor: Örebro University, Sweden (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: ORU 4.2-02319/2021; 2021-02653 (Other Grant/Funding Number: Swedish Research Council (Vetenskapsrådet))
Record Dates: First submitted 2025-05-07; First posted 2025-05-18 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Incontinence Associated Dermatitis
Keywords: Dermatitis; Risk factors; Urinary incontinence; Fecal incontinence; Prognosis
MeSH Terms: conditions — Dermatitis; Urinary Incontinence; Fecal Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Objective: The primary goal of this prospective cohort study is to collect data on specific factors, including age, sex, stool consistency, etc. and assess their association with the development of IAD. Through the compilation of this data, the study aims to determine whether the identified factors are indeed risk factors for the occurrence of IAD.

Study design: Prospective observational cohort study

Methodology:

This is a multi-center, prospective cohort study in hospitals in Sweden and Belgium. Adult patients (≥18 years) who are incontinent and free of IAD at baseline will be enrolled following informed consent.

Data collection: Daily skin assessments of the perineal area will be conducted by trained nurses using the validated Ghent Global Incontinence-Associated Dermatitis Tool (GLOBIAD). If IAD is detected, standardized photographs will be taken for blinded central review by skin integrity experts. Clinical, demographic, and care-related data will be collected, including variables such as age, sex, stool consistency, mobility, hygiene practices, nutrition, medication use, and comorbidities.

The primary endpoint for this study is to establish an association between the identified factors and the development of IAD in the study population.

DETAILED DESCRIPTION:
Problem Statement:

Incontinence-Associated Dermatitis (IAD) is a type of irritant contact dermatitis caused by prolonged skin exposure to urine and/or feces. It commonly affects individuals with incontinence. IAD is associated with decreased quality of life, increased care burden, loss of independence, and higher susceptibility to secondary infections and pressure ulcers. These complications lead to prolonged hospital stays and increased healthcare costs.

Despite its clinical relevance, there is insufficient consensus regarding the most critical risk factors for IAD. Existing literature points to a wide range of potential contributors including patient demographics, comorbidities, hygiene practices, and care protocols. A comprehensive prospective study is needed to investigate these risk factors within a hospitalized population in order to inform effective prevention and management strategies.

Methodology:

A prospective cohort design will be conducted across multiple hospital settings in Sweden and Belgium. The study targets adult patients, aged 18 years or older, who suffer from urinary, fecal, or double incontinence upon admission to the hospital and are free of IAD at enrollment.

The primary goal of this prospective cohort study is to collect data on specific factors, including age, sex, stool consistency, etc. and assess their association with the development of IAD. Through the compilation of this data, the study aims to determine whether the identified factors are indeed risk factors for the occurrence of IAD.

Data Collection:

Data collection will be managed through an electronic case report form (eCRF) using the RedCap® platform. Nurses will conduct daily inspections of the perianal skin area for each patient, recording observations and, when signs of IAD were identified, capture photographic evidence. These images will be reviewed by a blinded expert panel from the SCENTR team at Örebro University to confirm the diagnosis.

Collected variables include demographic data such as age, sex, and body weight, as well as clinical and care-related factors. These encompass comorbidities (e.g., diabetes, dermatological conditions, Clostridioides difficile infection), cognitive status, smoking habits, nutritional support (including enteral and parenteral nutrition), sedative and vasopressor use, and antibiotic therapy. Care-related variables include the frequency and type of incontinence, the number of absorbent product changes, skin cleansing and barrier product usage, and whether patients are mechanically ventilated. Additionally, functional assessments based on selected Braden Scale subscales-moisture, friction/shear, self-care ability, and mobility-will be recorded. Stool consistency will be classified using the Bristol Stool Chart, with a particular focus on types 6 and 7 (loose and watery stools), which have been previously identified as potential contributors to skin breakdown.

Data Analysis:

Statistical analysis, conducted using SPSS statistical package version 28.0 or later, will involve presenting summary statistics for demographics and clinical characteristics. Univariate analyses will explore associations between potential risk factors and IAD development, employing appropriate tests. Variables with p ≤ 0.2 significance in bivariate analysis will undergo multivariate logistic regression. Beforehand, multicollinearity will be assessed using multiple linear regression, and variables will be removed via the backwards method with P = 0.1 cut-off. Model fit will be evaluated using Nagelkerke R2 and Hosmer-Lemeshow statistic, with significance set at α = 0.05.

ELIGIBILITY:
Inclusion Criteria:

* The patient or their legally authorized representative signed informed consent.
* The patient is aged 18 years or older.
* The patient suffers from incontinence* (urinary, faecal, double incontinence).
* The patient is free of IAD at inclusion. *Incontinence is defined as involuntary loss of urine and/or stool.

Exclusion Criteria:

* Patients admitted to emergency departments, paediatric units, maternity units, psychiatric units, and palliative care units.
* Patients who are receiving end-of-life care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population includes adult hospitalised patients with urinary, faecal, or double incontinence who are free of IAD at inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 1037 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Association between prognostic factors and the development of IAD | 12 months
  This outcome will assess the relationship between selected prognostic factors (e.g., age, sex, stool consistency, type of incontinence) and the development of incontinence-associated dermatitis (IAD) in hospitalized incontinent patients. IAD status will be assessed using the GLOBIAD (Ghent Global IAD Categorisation Tool). The association between each prognostic factor and IAD will be evaluated using multivariable logistic regression analysis.

SECONDARY OUTCOMES:
Incidence of Incontinence-Associated Dermatitis (IAD) in hospitalized incontinent patients | 12 months (during the hospital stay of each enrolled patient, over the 12-month study period)
  The incidence of IAD will be measured as the proportion of hospitalized patients with urinary, fecal, or dual incontinence who develop IAD during their hospital stay. IAD will be assessed using the GLOBIAD (Ghent Global IAD Categorisation Tool).

CONTACTS AND LOCATIONS:
Overall Officials: Dimitri Beeckman, Professor, PhD, MSc, RN, Principal Investigator — Swedish Centre for Skin and Wound Research (SCENTR), School of Health Sciences, Faculty of Medicine and Health, Örebro University, Örebro, Sweden
Locations (7):
- Belgium (6):
  - AZ Sint-Lucas, Ghent
  - University Hospital Ghent, Ghent
  - Sint-Jozefskliniek, Izegem
  - AZ Groeninge, Kortrijk
  - AZ Delta, Rumbeke
  - AZ West, Veurne
- Uppsala University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deprez J, Kottner J, Eilegard Wallin A, Ohde N, Baath C, Hommel A, Hultin L, Josefson A, Beeckman D. What are the prognostic factors for the development of incontinence-associated dermatitis (IAD): a protocol for a systematic review and meta-analysis. BMJ Open. 2023 Jul 10;13(7):e073115. doi: 10.1136/bmjopen-2023-073115. PMID 37429690
- [Background] Deprez J, Ohde N, Eilegard Wallin A, Baath C, Hommel A, Hultin L, Josefson A, Kottner J, Beeckman D. Prognostic factors for the development of incontinence-associated dermatitis (IAD): A systematic review. Int Wound J. 2024 Jul;21(7):e14962. doi: 10.1111/iwj.14962. PMID 39016196